CLINICAL TRIAL: NCT00563693
Title: Open Randomized Study of Patients With Chronic Heart Failure and Cheyne Stokes Respiration Pattern, Treated With ASV. (Adaptive Servo Ventilator).
Brief Title: Chronic Heart Failure - Cheyne Stokes Respiration - CS2 (3C-study)
Acronym: 3C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Arild Hetland, MD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.2007.980
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure; Cheyne Stokes Respiration
Keywords: heart failure; cheyne stokes respiration; adaptive servo ventilator
MeSH Terms: conditions — Heart Failure; Cheyne-Stokes Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The patients use ASV
  Interventions: Device: ASV; Other: without Autoset CS2
- B (Active Comparator): Patients without ASV
  Interventions: Other: without Autoset CS2

INTERVENTIONS:
Device: ASV — Adaptive servo ventilator
  Other Names: AutoSet CS2
  Arms: A
Other: without Autoset CS2 — without Autoset CS2

SUMMARY:
An investigation where patients with chronic heart failure and cheyne stokes respiration, treated with adapitve servo ventilator, will improve their cardiac function and quality of life.

DETAILED DESCRIPTION:
Chronic heart failure (HF) is one of the most important public health problems in cardiovascular medicine.

Several patients with chronic heart failure also has Cheyne Stokes respiration pattern. Earlier studies have shown that this respiration pattern improves with Adaptive servo ventilator. We wish to investigate wether this leads to improved cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction <40%
* NYHA class III-IV
* Optimized therapy with drugs
* Cheyne stokes respiration pattern > 25% while sleeping
* Age < 85 years
* clinical stability the last month before inclusion.

Exclusion Criteria:

* CABG less then 6 months ago
* PCI treatment less then 3 months ago
* Unstable angina pectoris
* Acute coronary syndrome less then 3 months ago
* Stroke less then 6 weeks ago
* Thoracal myopathy
* Advanced COPD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Ejection fraction (measured with echocardiography) and inflammatory markers | 3 months

SECONDARY OUTCOMES:
6 minutes walking test Quality of life Changes in cathecolamines Altered frequency of arrythmias | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arild Hetland, cardiologist, Principal Investigator — University of Oslo
Locations (1):
- Sykehuset ostfold Fredrikstad, Fredrikstad, Norway